CLINICAL TRIAL: NCT04340739
Title: GEMINI: Virtual Integrative Medicine Group Visits (IMGV) for Managing Chronic Pain
Brief Title: Group intEgrative MINdfulness Over the Internet Using an Online Platform
Acronym: GEMINI
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); BrightOutcome (Industry)
Responsible Party: Principal Investigator, Paula Gardiner, Associate Professor, Associate Research Director, Medical Group Visit Program Director, University of Massachusetts, Worcester
Other Study IDs: H00017069; 1R43AT010460-01 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-04-09 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Pain, Chronic
Keywords: Widespread Chronic Pain; Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 (8 Patients): A wireframe mock-up of the GEMINI platform will be usability tested by 8 chronic pain patients from whom feedback will be collected by completing a virtual semi-structured interview. Outcomes: Quantitative Testing Data from Usability Testing Prompt. Qualitative data collected as feedback from semi-structured interview using the Usability Test Moderator Guide.
  Interventions: Other: online patient education teach mindfulness based stress reduction
- Cohort 2 (16 Patients): A live version of GEMINI will be beta-tested by 16 chronic pain patients through completing a faux medical group visit (MGV). This will include things like exploring the education topics available, interacting with the other participating patients, and interacting with a medical provider posing as the faux group's health care provider, all in order to robustly test the system in a "live" environment. Outcomes: Quantitative Testing/User Experience Data from Usability Testing Prompt, System Usability Scale, Perceived Feature Usefulness Scale, and the Technology Acceptance Model Based Survey. Qualitative data collected as feedback from semi-structured interview using the Usability Test Moderator Guide.
  Interventions: Other: online patient education teach mindfulness based stress reduction
- Cohort A (8 Healthcare Providers): Eight healthcare providers will be divided into pairs, and these pairs will each conduct a faux medical group visit (MGV) with faux patients (staff will pose as patients). They will be asked to complete the faux session as if it were actual patients of theirs, conduct pre- and post-session tasks, and provide usability feedback on the platform. Outcomes: Quantitative Testing/User Experience Data from Usability Testing Prompt, System Usability Scale, Perceived Feature Usefulness Scale, and the Technology Acceptance Model Based Survey. Qualitative data collected as feedback from semi-structured interview using the Usability Test Moderator Guide.
  Interventions: Other: online patient education teach mindfulness based stress reduction

INTERVENTIONS:
Other: online patient education teach mindfulness based stress reduction — This is an online self management chronic pain curriculum that presents adapted Mindfulness Based Stress Reduction through videos, audios, and written materials

SUMMARY:
This is a one-year study designed to improve upon the latest version of an education website for adult chronic pain patients called Our Whole Lives for Chronic Pain (OWL-CP). We will gain feedback from stakeholders, beta test new versions, and add the ability to conduct live Medical Group Visits through and on the virtual platform we are creating, GEMINI.

DETAILED DESCRIPTION:
The objectives are:

1. To create a wireframe version of the Group Integrative Mindfulness over the Internet (GEMINI) website, based on feedback from previous projects, for further beta testing.
2. To engage 8 patients with chronic pain in a focus group or individual meeting (utilizing the video-conferencing tool, Zoom) to obtain feedback on the wireframe version of GEMINI through a usability test and qualitative, semi-structured interview (Cohort 1).
3. To create a prototype of the GEMINI system, using all previously collected feedback data (mentioned above), for further beta testing with both patients and providers.
4. To engage 16 patients with chronic pain in focus group(s) to collect feedback on the patient portal side of the tool, through holding a non-intervention, GEMINI telehealth session using the prototype website. No personal health information (PHI) or medical record data will be collected or recorded during this faux session (Cohort 2).
5. To engage 8 health care providers in evaluating the provider portal through asking them to conduct a GEMINI telehealth session with study staff role-playing as chronic pain patients (Cohort A).
6. To end the project with a tested, active prototype of the GEMINI chronic pain management/education/telehealth tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older (Patients and Healthcare Providers (HCP))
* self-reported chronic physical pain for at least 12 weeks (Patients)
* average pain intensity for the previous week >4 on a 0 to 10 numerical rating scale (Patients)
* English fluency enough to follow instructions and answer survey questions (Patients and HCPs)
* Providers who treat patients for pain will be eligible for inclusion (HCPs)

Exclusion Criteria:

* Subjects who are not willing or unable to participate in a focus group or individual appointment over a video conferencing platform/on the University of Massachusetts (UMass) Worcester campus and watch a computer screen and give feedback (Patients

  * HCP)
* Fetuses, prisoners, and other vulnerable populations are not eligible (Patients & HCP)
* Providers/medical students or residents directly supervised by or reporting to the Primary Investigator (HCP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients will be recruited from the local Central Massachusetts area, with a focus on the adult primary care clinics within the UMass Memorial System. Providers can and will be recruited nationally through listservs, professional organizations, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Qualitative Feedback (Cohort 1) | Following 30 minute hands-on evaluation of system and brief (max 10 mins) survey collection (SUS, listed as add'l outcomes), duration of up to 1 hour. Session max of 2 hours.
  Prototype feedback collected during a 30 min to 1 hour semi-structured interview that will be held either in person or virtually, as able and with following all external guidelines.
Qualitative Feedback (Cohort 2) | Following 30 minute hands-on evaluation of system and brief (max 30 mins) survey collection (SUS, PFU, TAM-B, all listed as add'l outcomes), duration of up to 1 hour. Session max of 2 hours.
  Prototype feedback collected during a 30 min to 1 hour semi-structured interview that will be held either in person or virtually, as able and with following all external guidelines.
Qualitative Feedback (Cohort A) | Following 30 minute hands-on evaluation of system and brief (max 30 mins) survey collection (SUS, PFU, TAM-B, all listed as add'l outcomes), duration of up to 1 hour. Session max of 2 hours.
  Prototype feedback collected during a 30 min to 1 hour semi-structured interview that will be held either in person or virtually, as able and with following all external guidelines.
System Usability Scale (SUS) | Following 30 minute hands-on evaluation of system, up to 10 minutes, followed by Qualitative Feedback collection to end session. Session max of 2 hours.
  Prototype feedback data collected from all 3 cohorts using the System Usability Scale (SUS). The System Usability Scale is a 10 item survey, with each item ranked on a Likert scale ranging from 1-5, with a calculated score ranging from 0-100 (Subtracting 1 from each odd-numbered item's answer value and for each even-numbered question, subtracting their value from 5, summing both question sets, then multiplying the sum by 2.5). Average scores must fall at or above 70 to equate acceptable usability. Further information regarding scoring can be found by reading Bangor A, Kortum P, Miller J. Determining what individual SUS scores mean: adding an adjective rating scale. J Usability Studies. 2009;4(3):114-123.
Perceived Feature Usefulness Scale (PFU) | Following 30 minute hands-on evaluation of system, up to 10 minutes (30 mins for all 3 surveys), followed by Qualitative Feedback collection to end session. Session max of 2 hours.
  Prototype feedback data collected from Cohorts 2 and A using the Perceived Feature Usefulness Scale, a to-be designed 5-point Likert scale (from strongly disagree to strongly agree) survey. PFU cannot be fully designed before the system functions and the site structure are finalized because it would specifically ask the subject to rate the usefulness of each major system feature to guide our future product development plans. For instance, the statements could be "It is useful to view the profiles of my fellow patients in the group" or "It is useful to receive reminder emails about upcoming group sessions."
Technology Acceptance Based Model Survey | Following 30 minute hands-on evaluation of system, up to 10 minutes (30 mins for all 3 surveys), followed by Qualitative Feedback collection to end session. Session max of 2 hours.
  Prototype feedback data collected from Cohorts 2 and A using the Technology Acceptance Based Model Survey, a 5-point Likert scale survey. This survey will be based on the Technology Acceptance Model (TAM) that has been studied extensively to predict the actual use of health information technology (HIT) systems (Holden RJ, Karsh BT. The technology acceptance model: its past and its future in health care. J Biomed Inform. 2010;43(1):159-172). Key constructs include perceived usefulness (e.g., helpful in managing pain), perceived ease of use (e.g., easy to learn, session not too long), social influence (e.g., group effects), and perceived behavioral control (e.g., feasibility of videoconferencing).

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gardiner, MD MPH, Principal Investigator — University of Massachusetts, Worcester; Niina Haas, MA, Study Director — BrightOutcome
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
As this is not a clinical trial and the only data being collected is quantitative and qualitative feedback on our team's prototype chronic pain patient education and disease management platform, we do not plan to share any data at this time.

REFERENCES:
- [Background] Gardiner P, Dresner D, Barnett KG, Sadikova E, Saper R. Medical group visits: a feasibility study to manage patients with chronic pain in an underserved urban clinic. Glob Adv Health Med. 2014 Jul;3(4):20-6. doi: 10.7453/gahmj.2014.011. PMID 25105072